CLINICAL TRIAL: NCT06976476
Title: Prospective Randomized Phase II Study Evaluating Efficacy and Safety of IgPro20 as Infection Prophylaxis in Patients With Multiple Myeloma and Hypogammaglobulinemia Receiving Therapy With a Bispecific Monoclonal Antibody (BsAbs)
Brief Title: Study of IgPro20 to Prevent Infection in People With Multiple Myeloma and Hypogammaglobulinemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-137
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Hypogammaglobulinemia; Hypogammaglobulinemia, Acquired
Keywords: Multiple Myeloma; Hypogammaglobulinemia; IgPro20; Memorial Sloan Kettering Cancer Center; 24-137
MeSH Terms: conditions — Multiple Myeloma; Agammaglobulinemia; Common Variable Immunodeficiency | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants will only be observed
- Standard of Care + IGRT prophylaxis with IgPro20 (Experimental): Participants will receive IGRT prophylaxis with IgPro20 in addition to standard of care
  Interventions: Drug: IgPro20

INTERVENTIONS:
Drug: IgPro20 — Will be administered in addition to Standard of Care treatment. IgPro20 is intended for subcutaneous administration using an infusion pump
  Other Names: HIZENTRA
  Arms: Standard of Care + IGRT prophylaxis with IgPro20

SUMMARY:
The main purpose of this study is to see if IgPro20 can prevent infection in people with multiple myeloma (MM) who have hypogammaglobulinemia from receiving bispecific monoclonal antibodies (BsAbs).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMM receiving a commercially available bispecific antibody
* Received at least 1 but no more than 4 cycles of BsAb
* Males or females greater than or equal to 18 years old at the time of consent
* ECOG ≤ 3
* Life expectancy > 12 months

Exclusion Criteria:

* HSCT within 3 months before enrollment
* Planned CAR-T therapy in the next 6 months
* >1 major (deep-seated) infection within the preceding 3 months
* HIV infection, Active HCV, or Active HBV infection
* Pregnancy
* Neutrophils < 500 x 10^9 per mL, Platelets < 30 x 10^9 per mL
* History of cancer other than MM in the last 3 years requiring active chemotherapy or radiation
* Known reaction/allergy to IgG products
* Intracranial hemorrhage or embolic CVA in the last 6 months
* Hyperproteinemia
* Protein-losing enteropathy
* Creatinine Cl <30 ml/min
* Documented progression on BsAb
* Known history of Hyperprolinemia
* On current or previous IVIG (in the last 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2029-05-08 (Estimated); Study Completion 2029-05-08 (Estimated)

PRIMARY OUTCOMES:
Difference in overall infection rates between Standard of Care participants and participants receiving IgPro20 | 6 months
  To compare overall infection rates amongst (RR) multiple myeloma patients with hypogammaglobulinemia receiving subcutaneous immunoglobulin (IgPro20) to those in observational arm over a 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Shahid, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activity), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org